CLINICAL TRIAL: NCT00101309
Title: A Phase I Pilot Study of Tumor Cell - B Lymphoblastoid Cell Line Vaccination in Pediatric Subjects With Relapsed Ewing's Sarcoma and Neuroblastoma
Brief Title: Vaccine Therapy and Interleukin-2 in Treating Young Patients With Relapsed or Refractory Ewing's Sarcoma or Neuroblastoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Milton S. Hershey Medical Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000404366; PSCI-18990
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2007-11

CONDITIONS: Neuroblastoma; Sarcoma
Keywords: recurrent neuroblastoma; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor
MeSH Terms: conditions — Neuroblastoma; Sarcoma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — aldesleukin

INTERVENTIONS:
Biological: aldesleukin
Biological: autologous EBV-transformed B lymphoblastoid-tumor fusion cell vaccine
Biological: therapeutic autologous lymphocytes

SUMMARY:
RATIONALE: Vaccines made from a person's tumor cells and white blood cells may make the body build an effective immune response to kill tumor cells. Interleukin-2 (IL-2) may stimulate the white blood cells to kill tumor cells. Biological therapies, such as cellular adoptive immunotherapy, stimulate the immune system and stop tumor cells from growing. Giving vaccine therapy with IL-2 may be a more effective treatment for Ewing's sarcoma or neuroblastoma.

PURPOSE: This phase I trial is studying the side effects of vaccine therapy when given with IL-2 in treating young patients with relapsed or refractory Ewing's sarcoma or neuroblastoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the safety of vaccination comprising autologous tumor cells fused with Epstein-Barr virus-transformed B-lymphoblastoid cells followed by interleukin-2 (IL-2) in children with relapsed or refractory Ewing's sarcoma or neuroblastoma.
* Determine antitumor immunity by examining cell phenotype and function in patients treated with this vaccine and cytotoxic T lymphocytes (CTL).
* Determine the safety of CTL and IL-2 in these patients.

OUTLINE: This is a pilot study.

Tumor cells and blood cells are collected from patients and expanded in vitro. Tumor cells and Epstein-Barr virus-transformed B-lymphoblastoid cells (derived from blood cells) are fused together to produce the vaccine.

* Vaccination: Patients receive vaccine comprising autologous tumor cells fused with Epstein-Barr virus-transformed B-lymphoblastoid cells subcutaneously (SC) once on days 0, 14, and 28 and interleukin-2 (IL-2) SC twice daily on days 1-7, 15-21, and 29-35.
* Cytotoxic T lymphocytes (CTL): After vaccination, patients with evidence of antitumor immunity undergo leukapheresis to collect white blood cells for CTL expansion. Some of these patients then receive CTL IV once on days 0, 14, and 28 and IL-2 SC twice daily on days 1-7, 15-21, and 29-35.

Patients are followed weekly for 2 weeks, every 2 weeks for 1 month, monthly for 3 months, and then every 2 months for up to 1 year post-vaccination. Patients who receive CTL are also followed annually for survival.

PROJECTED ACCRUAL: A total of 10 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of Ewing's sarcoma OR neuroblastoma

  * Relapsed or refractory disease
* Epstein-Barr virus positive

PATIENT CHARACTERISTICS:

Age

* 1 to 30

Performance status

* Lansky 70-100% OR
* ECOG 0-2

Life expectancy

* At least 8 weeks

Hepatic

* Bilirubin < 2.0 mg/dL
* AST and ALT < 2.5 times normal (in the absence of liver metastases)

  * Patients without evidence of an obvious relationship between AST/ALT and disease activity are not eligible
* Hepatitis B antigen and core antibody negative
* Hepatitis C antibody negative

Renal

* Creatinine clearance > 50 mL/min

Immunologic

* HIV 1 and 2 negative
* HTLV 1 and 2 negative

Other

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other moribund condition

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 3 months since prior autologous stem cell transplantation

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 1 Year to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Estimated)
Dates: Start 2004-11; Primary Completion 2007-11 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth G. Lucas, MD, Study Chair — Milton S. Hershey Medical Center
Locations (1):
- Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States